CLINICAL TRIAL: NCT03652675
Title: Understanding and Intervening With Heavy Drinking Among Patients With HIV and HCV: Clinical Trial
Brief Title: Understanding and Intervening With Heavy Drinking Among Patients With HIV and HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jennifer C Elliott, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7649; K23AA023753 (NIH)
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Use Disorder; HIV/AIDS; Hepatitis C; Binge Drinking
Keywords: Heavy Drinking; HIV; Hepatitis C
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome; Hepatitis C; Binge Drinking | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After participants complete the screening assessment, the research coordinator will be able to determine alcohol use disorder status from the responses. The research coordinator will provide the counselor or PI with subject identification number (ID; assigned consecutively) and alcohol use disorder status. The counselor or PI will then randomize participants using pre-determined blocked lists created by a biostatistician, in order to balance treatment groups across alcohol use disorder status (the research coordinator will not randomize in order to remain blind to condition).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: (Clinician's Guide + HealthCall for HIV/HCV) (Experimental)
  Interventions: Behavioral: Intervention: (Clinician's Guide + HealthCall for HIV/HCV)
- Educational control condition (No Intervention): Participant will spend 20 minutes at the clinic, observed by the counselor, reviewing an educational pamphlet on drinking, HIV, and HCV.

INTERVENTIONS:
Behavioral: Intervention: (Clinician's Guide + HealthCall for HIV/HCV) — This intervention consists of an adaptation of the National Institutes of Health (NIH) Clinician's Guide (CG; NIAAA, 2007) in conjunction with the previously tested HealthCall smartphone app program (Hasin et al., 2013; Hasin et al., 2014). Participants will complete a brief baseline meeting (~20 minutes) with a counselor to discuss alcohol use, liver function, and HIV medication adherence. They will track their drinking using HealthCall for 60 days, with brief follow-up meetings with their counselor to check in about their drinking 30 and 60 days later.
  Arms: Intervention: (Clinician's Guide + HealthCall for HIV/HCV)

SUMMARY:
Among patients with HIV, especially those also infected with HCV, heavy drinking is associated with significant risks to health. However, little is known about how to best intervene with co-infected heavy drinkers, a particularly high risk group for whom targeted intervention has not been developed. Therefore, this study proposes to test a newly developed drinking-reduction intervention for patients with both HIV and HCV, which combines components of successful interventions developed for HIV and for liver disease patients.

60 HIV/HCV co-infected drinkers from HIV primary care will be recruited in order to ensure an adequate final sample size of 45 participants completing the study. A clinic recruiter will identify and refer potential participants based on their medical record, who will then be screened for eligibility by the research coordinator. Potential participants from outside of this clinic will also be recruited through self-referrals via flyers and through RecruitMe, an online based recruitment tool. Participants will be randomly assigned to an intervention or control condition, while ensuring that equal numbers of individuals with alcohol use disorder are assigned to each condition. The intervention condition will receive brief in-person sessions with a counselor and will be asked to use a smartphone app daily to keep track of drinking and other health behaviors for two months. The intervention sessions will include information about HIV, HCV and alcohol, and the counselor will give the participant information about their liver function and alcohol use to try to motivate them to drink less. The control condition will simply be asked to drink less and will be given pamphlets with general information on HIV, Hepatitis C, and drinking from educational websites on HIV/HCV co-infection. The intervention condition will then be evaluated to see if it was more effective at reducing drinking than the control condition.

DETAILED DESCRIPTION:
Patients with HIV have high rates of heavy drinking and alcohol problems, and face serious medical consequences from this use. Some research suggests that alcohol can increase viral load and decrease CD4 (cluster of differentiation 4; e.g., T helper cells) count, although this literature is conflicting. It also increases risk for liver damage, as does hepatitis co-infection, making liver disease a leading cause of death for patients with HIV. Patients with alcohol problems are also less adherent to antiretroviral therapy (ART), and some intentionally skip ART to try to avoid hepatotoxic effects of combining ART with alcohol. Some studies also show alcohol's interference with other aspects of engagement in HIV care.

Approximately 25% of HIV-infected patients are co-infected with HCV. Although HCV alone can lead to liver damage, HIV accelerates this progression, as does heavy drinking. Further, individuals with HCV who drink heavily may be less likely to access HCV medication. Despite serious health risks associated with alcohol use, some research suggests that HIV/HCV patients drink more than HIV mono-infected patients.

Growing recognition of alcohol-related harm in HIV patients has stimulated the development of drinking reduction interventions for HIV infected heavy drinkers, some of which have been successful. Some interventions for HCV mono-infected drinkers and liver disease patients have also shown promise. Yet there are no known successful interventions that target HIV/HCV co-infected patients, a group with elevated drinking and particularly high consequences of drinking. Interventions for HIV patients address HIV health, but do not address liver fibrosis, which is an urgent threat to survival for co-infected patients. Interventions for liver disease patients discuss fibrosis to motivate drinking reduction, but neglect HIV and important topics such as ART adherence. Given that the drinking interventions for HIV and liver disease patients both effectively target drinking in medical patients, albeit through attention to different medical issues, such approaches can and should be integrated to provide an intervention that best meets the needs of patients with both HIV and HCV, a particularly high-risk group. In order to meet this need, an intervention will be tested for HIV/HCV co-infected drinkers. A total of 60 patients will be recruited and randomized to receive either the newly developed intervention or an educational control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 99 (inclusive)
* HIV infection
* Ever been diagnosed with HCV infection (regardless of treatment status; including active or remitted infection)
* Recent (last 3 month) liver panel results available
* During prior 30 days, ≥4 drinks in one day at least once
* Can speak and read English
* Current and regular HIV care in NYC metro area

Exclusion Criteria:

* Participation in ongoing HealthCall study at Montefiore Hospital
* Potential participant has definite plans to leave the greater New York metropolitan area during study period
* Potential participant is psychotic, suicidal, or homicidal
* Potential participant is at-risk for developing alcohol withdrawal symptoms

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Elliott, Ph.D, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- NewYork-Presbyterian / Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasin DS, Aharonovich E, Greenstein E. HealthCall for the smartphone: technology enhancement of brief intervention in HIV alcohol dependent patients. Addict Sci Clin Pract. 2014 Feb 17;9(1):5. doi: 10.1186/1940-0640-9-5. PMID 24533631
- [Background] Hasin DS, Aharonovich E, O'Leary A, Greenstein E, Pavlicova M, Arunajadai S, Waxman R, Wainberg M, Helzer J, Johnston B. Reducing heavy drinking in HIV primary care: a randomized trial of brief intervention, with and without technological enhancement. Addiction. 2013 Jul;108(7):1230-40. doi: 10.1111/add.12127. Epub 2013 Apr 17. PMID 23432593
- See also: National Institute on Alcohol Abuse and Alcoholism - Helping Patients Who Drink Too Much: A Clinician's Guide — https://www.niaaa.nih.gov/guide

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Started | 16 | 15
Completed | 12 | 11
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (11.2) | 56.1 (9.7) | 56.4 (10.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12 | 9 | 21
  Female | 4 | 4 | 8
  Transgender | 0 | 1 | 1
  Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 31
Baseline Drinks per Drinking Day [Mean (Standard Deviation); unit: Drinks] | 5.24 (3.8) | 6.09 (2.17) | 5.65 (3.10)

OUTCOME MEASURES:

1. Primary Outcome: Mean Drinks Per Drinking Day Measured Using Timeline Follow Back (TLFB) at 60 Days.
Description: Mean drinks per drinking day in the last 30 days, assessed at baseline and repeatedly during follow-up so that change can be analyzed. Abstention is coded as zero.
Time Frame: 60 days (end of treatment)
Population: Of the 31 participants enrolled at baseline, 23 completed the 60-day follow-up and are reported here.
  Drinks per drinking day (primary outcome), with abstention coded as zero, at 60 days (end-of-treatment)
Measure: Mean (Standard Deviation); unit: Drinks per drinking day
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 11
Drinks per drinking day | 2.61 (3.35) | 5.49 (4.24)

2. Secondary Outcome: Change in Number of Days Drank as Assessed by Item From the Alcohol Use Disorder and Associated Disabilities Interview Schedule (AUDADIS)
Description: Number of days drank in the last 30 days (RANGE 0-30) was assessed at baseline and repeatedly during follow-up so that change can be analyzed. A change value is calculated here such that a negative value indicates a decrease in drinking.
Time Frame: 60 days (end of treatment)
Population: Of the 31 participants enrolled at baseline, 23 completed the 60-day follow-up and are reported here.
  Change scores from baseline - AUDADIS drinking variables at 60 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 11
Days | -6.08 (10.75) | -3.09 (10.4)

3. Other Pre Specified Outcome: Self-efficacy to Change Drinking as Measured by Brief Version of Situational Confidence Questionnaire (SCQ)
Description: Self-efficacy to change drinking in the last 30 days, assessed at baseline and repeatedly during follow-up so that change can be analyzed. Participants rate eight situations regarding their confidence in their ability to resist drinking (0% - Not at all confident to 100% - Totally confident). The final score is an average that can range from 0 (lowest) to 100 (highest) self-efficacy.
Time Frame: 60 days (end of treatment)
Population: Of the 31 participants enrolled at baseline, 23 completed the 60-day follow-up.Two participants were missing SCQ data at 60 days, so results are reported for 21 participants.
  Self-efficacy at 60 days (end-of-treatment), as measured by brief version of Situational Confidence Questionnaire (SCQ)
Measure: Mean (Standard Deviation); unit: Points on the SCQ
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 9
Points on the SCQ | 74.86 (17.99) | 66.3 (17.52)

4. Other Pre Specified Outcome: Readiness to Change Drinking Measured by University of Rhode Island Change Assessment Scale (URICA)
Description: Readiness to change drinking in the last 30 days, assessed at baseline and repeatedly during follow-up so that change can be analyzed.
  Higher scores indicate more readiness to change. Range from -2 to +14.
  The scale is scored when points are averaged for all four (precontemplation, contemplation, action, maintenance) scales. Add Contemplation + Action + Maintenance averages, then subtract Precontemplation average.
Time Frame: 60 days (end of treatment)
Population: Of the 31 participants enrolled at baseline, 23 completed the 60-day follow-up and are reported here.
  Readiness to change, as measured by the URICA
Measure: Mean (Standard Deviation); unit: Points on the URICA
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 11
Points on the URICA | 9.82 (2.16) | 8.98 (1.67)

5. Other Pre Specified Outcome: Readiness to Change Drinking Measured by The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES)
Description: Readiness to change drinking in the last 30 days,assessed at baseline and repeatedly during follow-up so that change can be analyzed.
  Higher scores indicate more recognition, ambivalence, and taking steps toward change, respectively. For full range and interpretation, see individual outcomes below.
  Recognition scale - Range 7 (very low recognition) to 35 (high recognition)
  Ambivalence scale - Range 4 (very low ambivalence) to 20 (very high ambivalence)
  Taking Steps scale - Range 8 (very low on taking steps to change drinking) to 40 (very high score)
Time Frame: 60 days (end of treatment)
Population: Of the 31 participants enrolled at baseline, 23 completed the 60-day follow-up and are reported here.
  SOCRATES subscales - Recognition, Ambivalence, Taking Steps
Measure: Mean (Standard Deviation); unit: Points on the SOCRATES subscales
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 11
Points on the SOCRATES subscales
  Recognition scale | 26.08 (6.4) | 26.55 (3.93)
  Ambivalence scale | 12.25 (2.99) | 13.36 (2.98)
  Taking Steps scale | 34.33 (4.79) | 28.73 (6.42)

6. Secondary Outcome: Change in Largest Number of Drinks Assessed by Item From the Alcohol Use Disorder and Associated Disabilities Interview Schedule (AUDADIS)
Description: The largest number of drinks consumed within one day in the last 30 days (RANGE 0-30) was assessed at baseline and repeatedly during follow-up so that change can be analyzed. A change value is calculated here such that a negative value indicates a decrease in drinking.
Time Frame: 60 days (end of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 11
drinks | -4 (5.15) | -5.36 (9.51)

7. Secondary Outcome: Change in Number of Days Binge Drinking as Assessed by Item From the Alcohol Use Disorder and Associated Disabilities Interview Schedule (AUDADIS)
Description: Number of days engaging in binge drinking (4+ drinks) in the last 30 days (RANGE 0-30) was assessed at baseline and repeatedly during follow-up so that change can be analyzed. A change value is calculated here such that a negative value indicates a decrease in drinking.
Time Frame: 60 days (end of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 11
days | -7.92 (8.24) | -6.27 (11.66)

8. Secondary Outcome: Change in Number of Days Intoxicated as Assessed by Item From the Alcohol Use Disorder and Associated Disabilities Interview Schedule (AUDADIS)
Description: Number of days intoxicated in the last 30 days (RANGE 0-30) was assessed at baseline and repeatedly during follow-up so that change can be analyzed. A change value is calculated here such that a negative value indicates a decrease in drinking.
Time Frame: 60 days (end of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
Number analyzed (Participants) | 12 | 11
days | -1.83 (4.13) | -0.64 (6.67)

ADVERSE EVENTS:
Time Frame: Every 30 days for 90 days.
Description: Consistent with ClinicalTrials.gov definition.
Arm/Group | Intervention: (Clinician's Guide + HealthCall for HIV/HCV) | Educational Control Condition
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

LIMITATIONS AND CAVEATS:
As recruitment started later and moved more slowly than intended, a smaller sample size than intended was obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03652675/Prot_001.pdf
  • Statistical Analysis Plan (2014-05-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03652675/SAP_002.pdf
  • Informed Consent Form (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03652675/ICF_000.pdf